CLINICAL TRIAL: NCT02768935
Title: Macrophage Phenotype in Type 2 Diabetics After Myocardial Infarction and the Potential Role of miRNAs Secreted
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOI-08
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: DIABETES; MYOCARD INFARCTUS
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes (Other)
  Interventions: Procedure: blood sample
- normoglycaemic (Other)
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — blodd sample at 12 months

SUMMARY:
The prevalence of type 2 diabetes is growing steadily. Patients with diabetes, cardiovascular complications (such as myocardial infarction (MI)) are more frequent and severe than in non-diabetic subjects. The anti-diabetic therapies available have little or no effect on the incidence of cardiovascular events. It is therefore urgent in diabetics develop new therapeutic strategies to reduce the occurrence of MI or limit the consequences.

In the two weeks following MI, monocytes / macrophages are the most represented in the ischemic heart tissue cells. The infiltration by monocytes / macrophages after infarction MI is a two-phase process. In the first phase, monocytes / macrophages M1 promote digestion injured areas, and monocytes / macrophages M2 intervene to promote angiogenesis, collagen deposition and contribute to tissue repair. The optimal repair after myocardial infarction depends on effective recruitment of monocytes and macrophages M1 transition needed to digest the damaged tissue and M2 macrophages necessary for tissue repair. The balance between these two phenotypes M1 and M2 is controlled by different modulators, such as transcription factors, cellular miRNA and miRNA extracellular contained in the microvesicles (MVs). Interestingly, plasma MVs circulating essentially derived monocytes and platelets contain miRNA and are impaired by inflammation or during various pathological situations (such as IDM). Furthermore, metabolic disorders such as hypercholesterolemia (often associated with diabetes) affect the transition from M1 to M2 response and response delay cardiac repair. To date, the mechanisms that control the M1 / M2 transition at heart level are not elucidated. Moreover, the impact of diabetes, which leads to chronic low-grade inflammation, is not explored. Targeting the immune response by promoting the transition M1 / M2 after MI could be an innovative therapeutic approach. However, better characterization of the response of M1 and M2 macrophages after MI and the mechanisms by which they contribute to tissue remodeling and the effect of diabetes are needed. The goal is to study how the phenotypes / macrophage functions after MI are changed by diabetes and to determine the potential role of miRNAs contained in secreted MVs in the transition M1 / M2 after MI.

Monocytes / macrophages from subjects with normal blood sugar or diabetes who underwent an IDM (10 per group) will be characterized phenotypically. Their ability to produce MVs will be analyzed. These MVs will be tested functionally for their ability to orient the polarization of healthy recipients monocytes. The content of these MVs in terms of miRNAs will be analyzed in detail. By bioinformatics analysis, some miRNAs of interest (based on their abundance and target genes) will be selected. These miRNAs are over-expressed in macrophages and MVs produced by these cells will be analyzed for their ability to modulate differentiation of monocytes recipients. Finally, the circulating levels of these miRNAs of interest will be measured after 1 year of IDM and will be correlated to the clinical phenotype of patients (recurrence, arrhythmias, heart failure). Ultimately, the goal is to identify VMs that can promote the differentiation of monocytes to an alternative phenotype and identify miRNAs responsible for this effect. This could help in the future, in a subject with impaired ability of monocytes to differentiate alternatively, can change by introducing the miRNA of interest to re-inject or inject MVs macrophage containing the miRNA of interest and thus correct the defect of differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Male Patients (to avoid the influence of estrogen hormones known to influence the M1 / M2 balance)
* Age: greater than 65 years (allowing homogeneity of the study population vis-à-vis the effect of age on differentiation M1 / M2)
* Patients hospitalized for a heart attack (chest pain, characteristic ECG changes, increased troponin levels (> 0.06 ng / ml))
* BMI between 19 and 30 (to avoid interference of obesity per se)
* Signed informed consent
* Affiliation to a social security scheme

Additional inclusion criterion for the group of diabetic subjects:

HbA1c of less than 2 months between 6 and 10% (to avoid confounding effects of anti-diabetic drugs).

Exclusion Criteria:

* Patients treated with anti-inflammatory agents (nonsteroidal anti-inflammatory drugs in the long term, corticosteroids, steroids, immunomodulators or immunosuppressants)
* Patients with acute inflammatory condition (in particular infectious)
* Patients with chronic inflammatory diseases (eg rheumatoid arthritis)
* Vulnerable Patients (convicts, under guardianship)

Ages: 65 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
level of expression markers | 12 months post myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No